CLINICAL TRIAL: NCT00150904
Title: Request for Blood Samples to Examine the Effect of Peginterferon and Ribavirin on Virologic and Immunologic Parameters in Patients With Hepatitis C and in Patients Coinfected With Hepatitis C and HIV
Brief Title: Peginterferon and Ribavirin on Virologic and Immunologic Parameters in Hepatitis C Mono- and Coinfected Patient (PRIVICOP)
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: 04-247E
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Hepatitis C; HIV Infections
Keywords: HIV; hepatitis C; virologic; immunologic; HIV / Hepatitis C coinfection
MeSH Terms: conditions — Hepatitis C; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: venous blood puncture

SUMMARY:
Hepatitis C and HIV infect worldwide millions of people leading to a high rate of coinfected patient with eventually liver cirrhosis and endstage liver disease. With the currently best available therapy (peginterferon and ribavirin) only less than 50% of patients with HCV genotype 1 will respond. Unknown is what factors determine this difference in treatment outcome. Probably virologic and immunologic factors play a major role. By investigating blood samples of HCV / HIV coinfected patients and HCV mono-infected patients we would like to examine both virologic and immunologic factors possibly responsible for this difference.

DETAILED DESCRIPTION:
background: each year the Hepatitis C (HCV) and the human immunodeficiency virus (HIV) infect worldwide millions of people. In the western world coinfection of HIV with HCV mainly exists in intravenous drug users. In coinfected patients progression of liver fibrosis to cirrhosis and endstage liver disease is much faster than in patients with only a mono-infection of hepatitis C. With the current treatment regimes response rates differ between HCV genotypes and between coinfected and mono-infected patients. Reasons for this a yet not well understood.

Virology: In the treatment of HCV genotype 1, after 12 weeks treatment success is evaluated (EVR) and if the HCV RNA-load is insufficiently dropped the treatment is stopped. There are indications that this moment of evaluation can be done earlier. Whole blood analysis can be a more sensitive method to determine an earlier EVR.Furthermore there are a few known HCV mutations playing a role in the chronicity of HCV. Lack of treatment response can be caused by other mutations in the HCV genome. Sequencing of the whole HCV genome has not been done very extensively.

Immunology: Proliferation and interferon production by HCV specific CD8 cells is defective. Not very much is known about the HCV-specific CD8 cells responses during treatment with peginterferon and ribavirin. Evidence is gathering that regulatory T-cells (CD4+CD25+) are involved in the process of inhibiting proliferation. Also it is known that the concentration of HCV-specific CD4 and CD8 cells in the liver is higher than in the peripheral blood. Certain homing molecules are probably involved in this process.

Hypothesis:

virologic: 1) at 4 weeks it is possible to determine an EVR; 2) other than the known ,mutations are responsible for the chronicity and unresponsiveness of the HCV virus; 3) whole blood analysis will be able to predict an EVR with more sensitivity than the current HCV-RNA techniques.

immunologic: 1) the specific relation between HCV specific CD4 and CD8 cells will determine if proliferation and production of interferon during therapy with peginterferon and ribavirin is successful. 2) regulatory T cells are inhibiting proliferation and production in chronic HCV infection and the amount of regulatory T cells will diminish during therapy with peginterferon and ribavirin. 3) wich homing molecules are important in the homing of HCV specific CD8 cells to the liver.

ELIGIBILITY:
Inclusion Criteria:

All patients where the treating physicians decides to start treatment with peginterferon and ribavirin for treatment of hepatitis C

* HCV mono-infection or HCV / HIV coinfection
* Genotype 1
* Compliant for outpatient visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I. M. Hoepelman, MD, PhD, Study Director — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Arends JE, Boucher CA, Hoepelman AI. Hepatitis C virus and human immunodeficiency virus coinfection: where do we stand? Neth J Med. 2005 May;63(5):156-63. PMID 15952483